CLINICAL TRIAL: NCT06092827
Title: Feasibility and Acceptability Study of a Non Weight-bearing Physical Activity Program for People With Diabetic Foot Ulceration (DB ACTIV)
Brief Title: Feasibility and Acceptability of Non Weight-bearing Physical Activity for People With Diabetic Foot Ulceration
Acronym: DB-ACTIV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Fondation Santé Trois-Rivières (Unknown); Centre intégré universitaire de santé et services sociaux Mauricie et Centre-du-Québec (CIUSSS MCQ) (Unknown); Université de Montréal (Other)
Responsible Party: Principal Investigator, Magali Brousseau-Foley, Principal Investigator, Université du Québec à Trois-Rivières
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F11-3298 : DB-ACTIV
Record Dates: First submitted 2023-01-16; First posted 2023-10-23 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot; Cardiopulmonary; Physical Inactivity
MeSH Terms: conditions — Diabetic Foot; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Feasibility and acceptability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical activity (Experimental): Adults 18 to 75 with an active diabetic foot ulcer
  Interventions: Behavioral: Non weight-bearing physical activity program

INTERVENTIONS:
Behavioral: Non weight-bearing physical activity program — 12-week duration, 2 supervised trainings/week, 1 unsupervised home-based training/week Aerobic, resistance and flexibility exercises

SUMMARY:
Intervention in the form of a PA (physical activity) program combining aerobic, resistance, and flexibility exercises adapted for wearing a lower limb offloading device and limiting weight-bearing on the feet, with a duration of twelve (12) weeks, consisting of two supervised sessions and one unsupervised home session per week.

DETAILED DESCRIPTION:
Objectives:

1. Evaluate the acceptability of a non-weight bearing physical activity (PA) program;
2. Assess the feasibility of the PA program and the data collection procedure;
3. Evaluate the feasibility of a submaximal exercise test for cardiorespiratory capacity; and
4. Verify the sensitivity of dependent variables to respond to a physical activity program (e.g., cardiorespiratory capacity, cardiovascular and metabolic risk factors, quality of life, PA level).

Type of study:

Feasibility and acceptability study with a pre-post evaluative design.

Intervention:

Intervention in the form of a PA (physical activity) program combining aerobic, resistance, and flexibility exercises adapted for wearing a lower limb offloading device and limiting weight-bearing on the feet, with a duration of twelve (12) weeks, consisting of two supervised sessions and one unsupervised home session per week.

Subjects:

* 10-12 persons with an active diabetic foot ulcer
* 2-3 kinesiologists

Data collection:

* Sociodemographic and health questionnaire (age, sex, gender, marital status, education level, employment status, average annual family income, medical and health history, pharmacological and non-pharmacological treatments);
* Feasibility assessment: PA (physical activity) logbook including 1) the number of supervised and unsupervised sessions completed, 2) the duration of each session, 3) participation rate (number of patients recruited/number of eligible patients), 4) attrition rate (number of participants who completed the follow-ups/number of participants recruited), and 5) perceived facilitators and barriers;
* Acceptability assessment: 1) Treatment Acceptability and Preference (TAP) Questionnaire, seven to nine additional questions to assess the use of provided material resources and required safety checks (capillary blood glucose and wound inspection) and collection of participants' feedback, and 2) Client Satisfaction Questionnaire (CSQ-8);
* Assessment of the sensitivity of dependent variables to respond to the PA program*: 1) estimation of VO2max by a submaximal exercise test on a stationary bike (Aerobic Power Index submaximal exercise test), 2) average daily step count over seven days at the waist and in the offloading boot at times 0, 4, 8, and 12 weeks, 3) Global Physical Activity Questionnaire (GPAQ), 3) clinical examination (height, weight, body mass index, waist circumference, body fat percentage, blood pressure, resting heart rate, characteristics of the DFU and classification (SINBAD), 4) paraclinical examinations (venous blood glucose, glycated hemoglobin, lipid profile), 5) neuropathic pain questionnaire (DN4), 6) Epworth sleepiness scale, quality of life questionnaire (EQ-5D-5L), 7) questionnaire on motivation to practice PA.
* Health and safety parameter measurements: electrocardiogram, oxygen saturation, estimated glomerular filtration rate, urine albumin/creatinine ratio, complete blood count.

  * Data collection at 24 and 36 weeks is also planned for participants who agree to be contacted after completing the 12-week PA program.

ELIGIBILITY:
For individuals with a diabetic foot ulcer:

Inclusion:

* Male or female
* Aged over 18 up to 75 years
* Willing to engage in PA (physical activity)
* Committed to following wound care recommendations to the best of their ability for the duration of the study
* Understand and read French.

Exclusion:

* Uncontrolled DFU infection
* Use of a non-removable offloading modality (total contact cast)
* Uncontrolled hyperglycemia (HbA1c ≥ 10.0% or fasting blood glucose ≥ 16.0 mmol/L for ≥ 2 consecutive days) confirmed by blood sample results during the initial assessment or access to recent blood test results (within the last 3 months) or the log of home capillary blood glucose readings
* Participation in sports or regular intense physical activities (≥ 2 times per week)
* The following pre-existing heart problems: a cardiovascular event (myocardial infarction, heart surgery, etc.) in the last 3 months, unstable cardiovascular disease (uncontrolled hypertension, i.e., ≥ 160/90 mmHg, uncompensated heart failure, etc.), chest pain and exertional dyspnea and/or uninvestigated intermittent claudication
* Recent neurovascular problem (stroke, transient ischemic attack, etc.) in the last 3 months
* Health problem that the research team considers a contraindication to participating in the study
* Diabetes complication making moderate-intensity PA unsafe, such as untreated proliferative diabetic retinopathy or a sensitivity disorder to hypoglycemia, critical ischemia of one or both lower limbs.

For kinesiologists:

Inclusion:

* Have completed a bachelor's degree in kinesiology
* Understand, read, and speak French.

Exclusion:

None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of physical activity intervention | At time 12 weeks
  Physical activity logbook, number of sessions completed with higher number meaning a greater feasibility
Acceptability of physical activity intervention | At time 12 weeks
  Treatment Acceptability and Preference (TAP) Questionnaire, minimum score 0/maximum score 16 with higher score meaning a greater acceptability
Satisfaction towards physical activity intervention | At time 12 weeks
  Client Satisfaction Questionnaire (CSQ-8), minimum score 8/maximum score 32 with higher score meaning a higher satisfaction

SECONDARY OUTCOMES:
Estimated VO2max | At times 0 and 12 weeks
  submaximal exercise test on a stationary bike (Aerobic Power Index submaximal exercise test), mL/kg/min
Average daily step count over seven days | At times 0, 4, 8, and 12 weeks
  At the waist and in the offloading boot using a FitBit Zip, number of steps
Physical activity level | At times 0 and 12 weeks
  Global Physical Activity Questionnaire (GPAQ), no minimum/maximum, details number of minutes/number of days per week of physical activity according to type of activity (work, leisures, commute, sedentary time)
Height | At time 0
  Standing with rigid measuring rod, cm
Weight | At times 0 and 12 weeks
  Standing on beam balance scale, kg
Waist circumference | At times 0 and 12 weeks
  With flexible measuring tape above ombilic, cm
Body fat percentage | At times 0 and 12 weeks
  With bio-impedance balance, %
Arterial blood pressure | At times 0 and 12 weeks
  With automatic blood pressure monitor, mm Hg
Resting heart rate | At times 0 and 12 weeks
  With automatic blood pressure monitor, bpm
Wound measurements (width, length, depth) | At times 0, 4, 8 and 12 weeks
  With flexible ruler
Classification of the ulcer | At times 0, 4, 8 and 12 weeks
  Using SINBAD system, 6 categories graded 0 or 1 for a minimum of 0 and maximum of 6, with higher score meaning a more complicated ulcer
Non fasting venous blood glucose | At times 0 and 12 weeks
  With venipuncture, mmol/L
Glycated hemoglobin | At times 0 and 12 weeks
  With venipuncture, %
Lipid profile (total cholesterol, low density lipoprotein, high density lipoprotein, triglycerides, non-HDL cholesterol) | At times 0 and 12 weeks
  Venipuncture, g/L
Neuropathic pain (if present) | At times 0 and 12 weeks
  Neuropathic pain (DN4) Questionnaire, 10 yes/no questions, higher number of yes indicates more severe neuropathic pain
Sleep apnea symptoms | At times 0 and 12 weeks
  Epworth sleepiness scale, minimum score of 0/maximum score of 24, higher score makes sleep apnea more likely
Reported quality of life | At times 0 and 12 weeks
  Quality of life questionnaire (EQ-5D-5L), minimum score of 5/maximum of 25 + 10cm visual analog scale, higher score represents a lower quality of life + 10cm being the best health condition possible
Questionnaire on motivation to practice physical activity | At times 0 and 12 weeks
  With the Behavioural Regulation in Exercise revised Questionnaire (BREQ-2), 5 motivation categories graded from 0 to 4, Intrinsic (4 questions), Identified (3 questions), Introjected (3 questions), External (4 questions) and Amotivation (4 questions), with lower scores meaning lesser motivation for each category

OTHER OUTCOMES:
Resting electrocardiogram (safety parameter) | At time 0
  To detect ST-T abnormalities at rest which has been shown to be most predictive for silent ischemia
Estimated glomerular filtration rate (safety parameter) | At times 0 and 12 weeks
  With venipuncture, mL/min. Results lower than 15 mL/min will need a specialist consultation to get medical clearance
Urine albumin/creatinine ratio (safety parameter) | At times 0 and 12 weeks
  With urinalysis, mg/g. Results lower than 300 mg/g will need a specialist consultation to get medical clearance
Hemoglobin (safety parameter) | At times 0 and 12 weeks
  With venipuncture, g/L. Results lower than 100 g/L will need a specialist consultation to get medical clearance

CONTACTS AND LOCATIONS:
Overall Officials: Magali Brousseau-Foley, MD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Universite du Quebec à Trois-Rivieres, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liubaoerjijin Y, Terada T, Fletcher K, Boule NG. Effect of aerobic exercise intensity on glycemic control in type 2 diabetes: a meta-analysis of head-to-head randomized trials. Acta Diabetol. 2016 Oct;53(5):769-81. doi: 10.1007/s00592-016-0870-0. Epub 2016 Jun 2. PMID 27255501
- [Background] Umpierre D, Ribeiro PA, Schaan BD, Ribeiro JP. Volume of supervised exercise training impacts glycaemic control in patients with type 2 diabetes: a systematic review with meta-regression analysis. Diabetologia. 2013 Feb;56(2):242-51. doi: 10.1007/s00125-012-2774-z. Epub 2012 Nov 16. PMID 23160642
- [Background] Umpierre D, Ribeiro PA, Kramer CK, Leitao CB, Zucatti AT, Azevedo MJ, Gross JL, Ribeiro JP, Schaan BD. Physical activity advice only or structured exercise training and association with HbA1c levels in type 2 diabetes: a systematic review and meta-analysis. JAMA. 2011 May 4;305(17):1790-9. doi: 10.1001/jama.2011.576. PMID 21540423
- [Background] Balducci S, Zanuso S, Cardelli P, Salvi L, Bazuro A, Pugliese L, Maccora C, Iacobini C, Conti FG, Nicolucci A, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Effect of high- versus low-intensity supervised aerobic and resistance training on modifiable cardiovascular risk factors in type 2 diabetes; the Italian Diabetes and Exercise Study (IDES). PLoS One. 2012;7(11):e49297. doi: 10.1371/journal.pone.0049297. Epub 2012 Nov 21. PMID 23185314
- [Background] Chudyk A, Petrella RJ. Effects of exercise on cardiovascular risk factors in type 2 diabetes: a meta-analysis. Diabetes Care. 2011 May;34(5):1228-37. doi: 10.2337/dc10-1881. PMID 21525503
- [Background] Cai H, Li G, Zhang P, Xu D, Chen L. Effect of exercise on the quality of life in type 2 diabetes mellitus: a systematic review. Qual Life Res. 2017 Mar;26(3):515-530. doi: 10.1007/s11136-016-1481-5. Epub 2016 Dec 18. PMID 27990609
- [Background] Nielsen PJ, Hafdahl AR, Conn VS, Lemaster JW, Brown SA. Meta-analysis of the effect of exercise interventions on fitness outcomes among adults with type 1 and type 2 diabetes. Diabetes Res Clin Pract. 2006 Nov;74(2):111-20. doi: 10.1016/j.diabres.2006.03.033. Epub 2006 Jun 2. PMID 16735074
- [Background] Wei M, Gibbons LW, Kampert JB, Nichaman MZ, Blair SN. Low cardiorespiratory fitness and physical inactivity as predictors of mortality in men with type 2 diabetes. Ann Intern Med. 2000 Apr 18;132(8):605-11. doi: 10.7326/0003-4819-132-8-200004180-00002. PMID 10766678
- [Background] Schaper NC, van Netten JJ, Apelqvist J, Bus SA, Hinchliffe RJ, Lipsky BA; IWGDF Editorial Board. Practical Guidelines on the prevention and management of diabetic foot disease (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3266. doi: 10.1002/dmrr.3266. PMID 32176447
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] Agence de la santé publique du Canada (ASPC). Le diabète au Canada : Perspective de santé publique sur les faits et chiffres 2011 [Available from: https://www.canada.ca/fr/sante-publique/services/maladies-chroniques/rapports-publications/diabete/diabete-canada-perspective-sante-publique-faits-chiffres.html.
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] van Netten JJ, Price PE, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Bus SA; International Working Group on the Diabetic Foot. Prevention of foot ulcers in the at-risk patient with diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:84-98. doi: 10.1002/dmrr.2701. PMID 26340966
- [Background] Ribu L, Hanestad BR, Moum T, Birkeland K, Rustoen T. A comparison of the health-related quality of life in patients with diabetic foot ulcers, with a diabetes group and a nondiabetes group from the general population. Qual Life Res. 2007 Mar;16(2):179-89. doi: 10.1007/s11136-006-0031-y. Epub 2006 Nov 8. PMID 17091370
- [Background] Hopkins RB, Burke N, Harlock J, Jegathisawaran J, Goeree R. Economic burden of illness associated with diabetic foot ulcers in Canada. BMC Health Serv Res. 2015 Jan 22;15:13. doi: 10.1186/s12913-015-0687-5. PMID 25608648
- [Background] Bissonnette V. Évaluation des coûts et éléments d'efficacité du traitement d'un ulcère du pied diabétique [Mémoire de maîtrise]: Université de Sherbrooke; 2011.
- [Background] Pelletier C, Dai S, Roberts KC, Bienek A, Onysko J, Pelletier L. Report summary. Diabetes in Canada: facts and figures from a public health perspective. Chronic Dis Inj Can. 2012 Dec;33(1):53-4. PMID 23294922
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Wallman K, Goodman C, Morton A, Grove R, Dawson B. Test-retest reliability of the aerobic power index component of the tri-level fitness profile in a sedentary population. J Sci Med Sport. 2003 Dec;6(4):443-54. doi: 10.1016/s1440-2440(03)80270-0. PMID 14723394
- [Background] Wallman KE, Campbell L. Test-retest reliability of the Aerobic Power Index submaximal exercise test in an obese population. J Sci Med Sport. 2007 Jun;10(3):141-6. doi: 10.1016/j.jsams.2006.05.024. Epub 2006 Jul 17. PMID 16844410
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Sigal RJ, Armstrong MJ, Bacon SL, Boule NG, Dasgupta K, Kenny GP, Riddell MC. Physical Activity and Diabetes. Can J Diabetes. 2018 Apr;42 Suppl 1:S54-S63. doi: 10.1016/j.jcjd.2017.10.008. No abstract available. PMID 29650112
- [Background] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Background] Borg G. Borg's perceived exertion and pain scales: Human kinetics; 1998.
- [Background] Thakur A, Sharma R, Sharma SK, Thakur K, Jelly P. Effect of buerger allen exercise on foot perfusion among patient with diabetes mellitus: A systematic review & meta-analysis. Diabetes Metab Syndr. 2022 Feb;16(2):102393. doi: 10.1016/j.dsx.2022.102393. Epub 2022 Jan 13. PMID 35085917
- [Background] Sidani S, Epstein DR, Bootzin RR, Moritz P, Miranda J. Assessment of preferences for treatment: validation of a measure. Res Nurs Health. 2009 Aug;32(4):419-31. doi: 10.1002/nur.20329. PMID 19434647
- [Background] Evenson KR, Goto MM, Furberg RD. Systematic review of the validity and reliability of consumer-wearable activity trackers. Int J Behav Nutr Phys Act. 2015 Dec 18;12:159. doi: 10.1186/s12966-015-0314-1. PMID 26684758
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Sabourin S, Pérusse D, Gendreau P. Les qualités psychométriques de la version canadienne-française du Questionnaire de Satisfaction du Consommateur de services psychothérapeutiques (QSC-8 et QSC-18B). Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement. 1989;21(2):147.
- [Background] Crews RT, Armstrong DG, Boulton AJ. A method for assessing off-loading compliance. J Am Podiatr Med Assoc. 2009 Mar-Apr;99(2):100-3. doi: 10.7547/0980100. PMID 19299344
- [Background] Armstrong T, Bull F. Development of the world health organization global physical activity questionnaire (GPAQ). Journal of Public Health. 2006;14:66-70.
- [Background] Fernandez-Torres R, Ruiz-Munoz M, Perez-Panero AJ, Garcia-Romero JC, Gonzalez-Sanchez M. Clinician Assessment Tools for Patients with Diabetic Foot Disease: A Systematic Review. J Clin Med. 2020 May 15;9(5):1487. doi: 10.3390/jcm9051487. PMID 32429068
- [Background] Spallone V, Morganti R, D'Amato C, Greco C, Cacciotti L, Marfia GA. Validation of DN4 as a screening tool for neuropathic pain in painful diabetic polyneuropathy. Diabet Med. 2012 May;29(5):578-85. doi: 10.1111/j.1464-5491.2011.03500.x. PMID 22023377
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Matza LS, Boye KS, Stewart KD, Curtis BH, Reaney M, Landrian AS. A qualitative examination of the content validity of the EQ-5D-5L in patients with type 2 diabetes. Health Qual Life Outcomes. 2015 Dec 1;13:192. doi: 10.1186/s12955-015-0373-7. PMID 26627874
- [Background] Ferrari M, Speight J, Beath A, Browne JL, Mosely K. The information-motivation-behavioral skills model explains physical activity levels for adults with type 2 diabetes across all weight classes. Psychol Health Med. 2021 Mar;26(3):381-394. doi: 10.1080/13548506.2020.1749292. Epub 2020 Apr 8. PMID 32266821